CLINICAL TRIAL: NCT01372358
Title: Single Dose, Randomized, Two-period, Two-treatment, Two-sequence Crossover Relative Bioavailability Study of Ciprofloxacin 1000 mg ER Tablets Under Non-Fasting Condition.
Brief Title: Bioavailability Study of Ciprofloxacin 1000 mg ER Tablets of Dr. Reddy's Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. M.S. Mohan/Vice President - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B045908
Record Dates: First submitted 2011-01-26; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-01

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin (Experimental): Ciprofloxacin Extended Release Tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: CIPRO®XR
- CIPRO®XR (Active Comparator): CIPRO® XR (Bayer Health Care, Bayer Pharmaceuticals Corporation) Tablets
  Interventions: Drug: CIPRO®XR

INTERVENTIONS:
Drug: CIPRO®XR — Ciprofloxacin 1000 mg Tablets Dr. Reddy's Laboratories Limited
  Other Names: CIPRO®XR tablets of Bayer Health Care

SUMMARY:
The purpose of this study is to compare the relative bioavailability of ciprofloxacin 1000 mg ER tablets of Dr.Reddy's with that of CIPRO® XR 1000 mg of Bayer Pharmaceuticals Corporation in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
This single dose, randomized, two-period, two-treatment, two sequence crossover study was conducted to compare the relative bioavailability of ciprofloxacin 1000 mg ER tablets of Dr. Reddy's and CIPRO® XR 1000 mg of Bayer Pharmaceuticals Corporation under non-fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Non-institutionalized subjects consisting of members of, the coInmunity at large.
2. All subjects selected for this study will be non-smokers between 18 and 45 years of age (inclusive). Female subjects must be unable to become pregnant (postmenopausal for at least 1 year, or surgically sterile)
3. Each subject shall be given, a general physical examination within 28 days of initiation of the study and will include, but is not limited to, blood pressure, general observations, and history.
4. Each female subject will be given a serum pregnancy test as part of the pre-study screening process.
5. Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.
6. Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

1. Subjects with a history of alcoholism or drug addiction (during past 2 years), or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
2. Subjects whose clinical laboratory test values are outside the normal range may be retested at the discretion of the clinical investigator. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
3. Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
4. All subjects will have urine / saliva samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at check-in each dosing period. Subjects found to have urine/saliva concentrations of any of the tested drugs will not be allowed to participate.
5. Subjects should not have donated blood and / or plasma for at least thirty (30) days prior to tile first dosing of the study.
6. Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
7. Female subjects who are pregnant or who are able (women with childbearing potential) to become pregnant during the study will not be allowed to participate.
8. All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
9. Subjects who have a history of clinically significant illnesses or surgery within 4 weeks prior to the administration of the study medication will not be eligible for this study.
10. Subjects who have a BMI ≥30.0 Kg/m2 will not be eligible for this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Saran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services, 3320 Walnut Bend Lane, Houston, Texas 77042-4712, United States of America (USA)
Locations (1):
- NOVUM Pharmaceutical Research Services, Houston, Texas, United States